CLINICAL TRIAL: NCT07343726
Title: Impact of Obesity on Response to Therapy and Clinical Outcom in Patients With Inflammatory Bowel Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Ahmed Mahmoud Abdelmohsen, residant doctor at Assiut university hospital, Assiut University
Other Study IDs: obesity IBS
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Inflammatory Bowel Disease (IBD)
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- obese patients: obese patients who have BMI ≥ 30
- non-obese patients: non-obese patients who have BMI < 30

SUMMARY:
Inflammatory Bowel Disease (IBD), which includes ulcerative colitis (UC) and Crohn's disease (CD), is a group of chronic relapsing inflammatory disorders of the gastrointestinal tract. Its pathogenesis is multifactorial, involving genetic predisposition, environmental triggers, immune dysregulation, and microbial imbalance. IBD has significant morbidity and a major impact on quality of life, with varied clinical presentations and disease behavior (1,2).

Obesity, defined as excessive body fat accumulation, is increasingly prevalent worldwide. It is now recognized as a state of chronic low-grade systemic inflammation due to adipose tissue secreting pro-inflammatory cytokines such as TNF-α and IL-6 (3,4). These cytokines may interact with pathways relevant to IBD, particularly in altering the immune response and intestinal inflammation (5).

recent studies suggest that obese IBD patients may experience a different disease phenotype, increased complications, and lower response rates to certain biologics, especially anti-TNF agents (6,7). In addition, obesity can alter drug pharmacokinetics, leading to reduced drug efficacy (8,9).

Despite increasing evidence of this association, there is limited local data evaluating the prevalence of obesity in IBD and its impact on treatment response and disease outcome (10,11). Understanding this link could help improve personalized treatment approaches and predict treatment outcomes in IBD patients (12,13).

Obesity has emerged as a modifiable factor that may influence the clinical response to therapy in patients with inflammatory bowel disease (IBD). Recent studies have shown that higher body mass index (BMI) is associated with reduced steroid-free clinical remission rates in patients treated with advanced biologic and small molecule therapies. The inflammatory nature of adipose tissue, altered pharmacokinetics, and increased drug clearance in obese individuals might explain the suboptimal therapeutic outcomes observed in this population

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years) diagnosed with IBD
* Currently receiving standard treatment (including biologics)

Exclusion Criteria:

* Patients with other causes of colitis (e.g. infectious, ischemic)
* Pregnant females
* Incomplete clinical or follow-up data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (>18 years) diagnosed with IBD
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
improvement rate of patients | 3 months
  Clinical response to treatment